CLINICAL TRIAL: NCT04104997
Title: A Randomized, Double-blind, Placebo-controlled Phase 1 Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of GLH8NDE After Single and Mutiple Ocular Administrations in Healthy Korean and Caucasian Volunteers
Brief Title: A Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of GLH8NDE After Single and Mutiple Ocular Administrations in Healthy Korean and Caucasian Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GLH8NDE-101
Record Dates: First submitted 2019-09-20; First posted 2019-09-26 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- The A group in 5% GLH8NDE (Experimental): Three times administration both eyes, each 1 drop in Korean
  Interventions: Drug: 5% GLH8NDE
- The A group in placebo (Placebo Comparator): Three times administration both eyes, each 1 drop in Korean
  Interventions: Drug: Placebos
- The B group in 5% GLH8NDE (Experimental): Six administration both eyes, each 1 drop in Korean
  Interventions: Drug: 5% GLH8NDE
- The B group in placebo (Placebo Comparator): Six administration both eyes, each 1 drop in Korean
  Interventions: Drug: Placebos
- The C group in 5% GLH8NDE (Experimental): Six administration both eyes, each 2 drop in Korean
  Interventions: Drug: 5% GLH8NDE
- The C group in placebo (Placebo Comparator): Six administration both eyes, each 2 drop in Korean
  Interventions: Drug: Placebos
- The D group in 5% GLH8NDE (Experimental): Six administration both eyes, each 2 drop in Caucasian
  Interventions: Drug: 5% GLH8NDE
- The D group in placebo (Placebo Comparator): Six administration both eyes, each 2 drop in Caucasian
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: 5% GLH8NDE — 5% GLH8NDE as eye drops
  Arms: The A group in 5% GLH8NDE; The B group in 5% GLH8NDE; The C group in 5% GLH8NDE; The D group in 5% GLH8NDE
Drug: Placebos — Placebo as eye drops
  Arms: The A group in placebo; The B group in placebo; The C group in placebo; The D group in placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled phase 1 clinical trial to evaluate the safety, tolerability and pharmacokinetic characteristics of GLH8NDE after single and multiple ocular administrations in healthy Korean and Caucasian volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject who, at the time of screening, are the age between 20 and 50 years
* Subject who has body weight between 55.0 and 90.0 kg, and BMI between 18.0 and 27.0
* Subject who signed and dated the informed consent form after understanding fully to hear a detailed explanation in the clinical trial

Exclusion Criteria:

* A subject who has a evidence or history of clinically significant hepatic, renal, neurologic, pulmonary, endocrine, urological, psychiatric, cardiovascular, hematological, oncological, etc.
* A subject who has a history of disease with myocardial infarction, stroke, arrhythmia, hypotension (90 mmHg amine or diastolic blood pressure less than 50 mmHg at screening), uncontrolled hypertension (greater than 170 mmHg diastolic blood pressure or 100 mmHg diastolic blood pressure at screening), coronary artery, or who has a current abnormality
* A subject with a history of hypersensitivity to the drug (aspirin, antibiotics, etc.) or clinical significant hypersensitivity reactions
* A subject with the following findings in paperweight, visual acuity test, front eye photo, corneal refraction test, intraocular pressure test, slit lamp microscopy examination, fundus examination, tear break-up time examination, tear secretion test, OSDI (ocular surface disease index) are excluded

  1. A subject with suspected history or symptoms of visual organs, including keratitis, uveitis, retinitis, dry eye and strabismus
  2. A subject who has had eye surgery (including those who have received more than 6 months for eye laser surgery)
  3. A subject at least one eye with an intra-ocular pressure of 22 mmHg or more at the screening
  4. At the screening, tear break-up time of at least one eye in both eyes is less than 10 seconds and diagnosed as dry eye according to OSDI test
  5. A subject whose ratio for at least one eye in both eyes during screening is less than 10 mm as measured for 5 minutes in an Un-anesthetized Schirmer's test
  6. There are side effects to people who wear contact lenses after wearing them or within a month
* A subject with a history of drug abuse or a positive urine drug screening for drug abuse
* A subject who has participated in any other clinical trials and bioequivalence had medication within 6 months prior to the first administration of investigational product (The end date of another clinical trial is based on the last day of the administration)
* A subject who has taken any ethical-the-counter drug or herbal drug within 2 weeks has taken any over-the-counter drug or vitamin include artificial tears within 1 week before the investigational product
* A subject who has donated whole blood within 2 months or blood components within 1 month prior to the investigational product administration
* History of regular alcohol consumption exceeding 21 units/week (1 unit = 10 g of pure alcohol) within 60 days before the investigational product or non-stop the alcohol drinking
* The current smoker, but except the subject to quit the smoke over 90 days
* Recognized contraceptive methods (e.g. your and your partner's infertility surgery, your partner's intrauterine device (IUD), cervical caps or contraceptive diaphragms for use with spermicides) Single block), cervical cap or contraceptive diaphragm with male condom (double block)]
* A subject who have to work that cause excessive eye fatigue during this clinical trial
* A subject who is not eligible for the study due to reasons on the investigators' judgement

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Adverse events | Between 1 day before first IP administration and 18 days
  To 18 days after first IP administration
Vital signs in blood pressure | Each point at Screening(between 2 day and 28 day before IP administration), 1, 2, 4, 6, 8, 10, 11 days, and post-study visit(between 16 and 18 days)
  Whether out of normal range at Blood pressure (SBP, DBP)
Vital signs in pulse | Each point at Screening(between 2 day and 28 day before IP administration), 1, 2, 4, 6, 8, 10, 11 days, and post-study visit(between 16 and 18 days)
  Whether out of normal range at Pulse rate
Vital signs in temperature | Each point at Screening(between 2 day and 28 day before IP administration), 1, 2, 4, 6, 8, 10, 11 days, and post-study visit(between 16 and 18 days)
  Whether out of normal range in temperature at eardrum
Physical examinations in weight change | Change trend of the each point among screening(between 2 day and 28 day before IP administration), 1, 2, 4, 6, 8, 10, 11 days, and post-study visit(between 16 and 18 days)
  Weight change in kilograms
Clinical laboratories in blood sample | Each point at day 1, 2, 4, 6, 8, 10, and 11
  Whether abnormal blood chemistry
Clinical laboratories in blood sample | Each point at day 1, 2, 4, 6, 8, 10, and 11
  Whether positive at Type B hepatitis, Type C hepatitis, HIV, and Syphilis
12-lead ECG in clinical significance | Each point at Screening(between 2 day and 28 day before IP administration), 1, 4, 11 days, and post-study visit(between 16 and 18 days)
  Whether out of normal range QRS complex
Ophthalmic symptom | Each point at Day 1, 2, 4, 6, 8, 10, and 11
  To 18 days after first IP administration
Ophthalmic examination | Each point at Screening(between 2 day and 28 day before IP administration), 2, 11 days, and post-study visit(between 16 and 18 days)
  Tear break-up time examination
AUClast in ng·h/mL | Pre-dose, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours after last administration
  One day administration as GLH8NDE
AUCinf in ng·h/mL | Pre-dose, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours after last administration
  One day administration as GLH8NDE
Cmax in ng/mL | Pre-dose, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours after last administration
  One day administration as GLH8NDE
Tmax in ng/mL | Pre-dose, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours after last administration
  One day administration as GLH8NDE
t1/2 in hour | Pre-dose, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours after last administration
  One day administration as GLH8NDE
AUCtau,ss in ng·h/mL | Pre-dose, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours after last administration
  Mutiple dose administration as GLH8NDE
Cmax in ng/mL | Pre-dose, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours after last administration
  Mutiple dose administration as GLH8NDE
Tmax in ng/mL | Pre-dose, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours after last administration
  Mutiple dose administration as GLH8NDE
t1/2 in hour | Pre-dose, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours after last administration
  Mutiple dose administration as GLH8NDE
R(Accumulation index) | Pre-dose, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours after last administration
  Accumulation in dex at mutiple dose administration as GLH8NDE

CONTACTS AND LOCATIONS:
Overall Officials: MinChang Kwon, Ph. D, Study Director — GL PharmTech Corp.
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea